CLINICAL TRIAL: NCT00221416
Title: An Open-Label Trial of Aripiprazole in Children and Adolescents With Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Robert Kowatch, Principal Investigator, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-7-11
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Bipolar Disorder
Keywords: child; adolescent
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aripiprazole — 5-20 mg/day

SUMMARY:
This is an investigator-initiated study whose primary aim is to determine the effectiveness of aripiprazole (Abilify®) in helping persons with symptoms of mania whose current medications do not completely control those symptoms. Aripiprazole is a medication that has been approved by the United States Food and Drug Administration (FDA) for the treatment of Schizophrenia.

A secondary aim of this research is to explore whether CYP 2D6 polymorphisms are related to side effects with aripiprazole. The goal of this research is to identify individuals who metabolize aripiprazole more rapidly or slowly, which will potentially help the clinician make dosing adjustments and decrease the risk of adverse events.

DETAILED DESCRIPTION:
The primary aim of this study is to assess the effectiveness, safety, and tolerability of aripiprazole for the treatment of children and adolescents with bipolar disorder. The secondary aim of this study is to determine if common polymorphic variations in the CYP 2D6 gene underlie the inter-individual variability in aripiprazole systemic drug exposure and the occurrence of treatment emergent side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Females; between the ages of 7 years 0 months to 17 years 12 months
2. Bipolar I Disorder, mixed or manic episode, psychotic or non-psychotic, according to DSM IV criteria.
3. Score of > 20 on the Y-MRS at baseline.
4. Ability and willingness to provide assent and informed written consent from at least one parent or legal guardian
5. No current general medical illnesses requiring medication that would effect interpretation of study outcomes.
6. Subjects must have at least normal intelligence.
7. Female patients of childbearing potential must be using a reliable method of contraception, e.g. hormonal contraceptives, Depo-Provera, double-barrier methods (e.g. condom and diaphragm, condom and foam, condom and sponge) or abstinence). Females of childbearing potential must have a negative serum pregnancy test immediately prior to study entry.
8. Must be able to swallow oral medication (tablets).

Exclusion Criteria:

1. A current or lifetime DSM-IV diagnosis of schizophrenia, autistic disorder, schizoaffective disorder, pervasive developmental disorder, or obsessive compulsive disorder
2. Known IQ < 70
3. Patients with high suicide risk defined as any serious suicide attempt that required medical intervention or current suicide risk that cannot be safely managed as determined by the clinical judgment of the investigator.
4. Concurrent cognitive behavioral psychotherapy.
5. Present or past (within 3 months) DSM-IV diagnosis of substance abuse/dependence.
6. Female patients who are pregnant, trying to become pregnant, nursing an infant, or not using a reliable form of contraception.
7. Bipolar subjects who are currently stable on mood stabilizers or atypical neuroleptics.
8. Patient has failed on a previous adequate course of aripiprazole.
9. A known hypersensitivity to aripiprazole or to any of its components.
10. Participated in an investigational drug/device trial within the last 30 days.
11. Patients with severe renal insufficiency, defined as creatinine clearance <30ml/min. by history or by lab findings.

    -

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
YMRS & CGI | 6 weeks

SECONDARY OUTCOMES:
OAS CDRS-R | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Kowatch, MD, Principal Investigator — University of Cincinnati